CLINICAL TRIAL: NCT00337220
Title: Noninvasive Diagnosis of Renal Allograft Rejection by Urinary Cell mRNA Profiling
Brief Title: Urine Testing to Detect Kidney Transplant Rejection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-04
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Kidney Transplantation; Kidney Disease; Kidney Failure, Chronic
Keywords: allograft; graft
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine collection
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if analysis of urine samples for specific markers can predict transplant rejection in people who have received kidney transplants.

DETAILED DESCRIPTION:
Innovations in kidney transplantation have improved short-term outcomes for transplant patients. However, organ rejection remains as an important threat to the long-term survival of the transplanted organ. An increase in the serum creatinine level is often the first clinical indicator of kidney transplant rejection; however, this marker lacks sensitivity and specificity. Rejection is currently diagnosed using an invasive transplant biopsy procedure; in addition to being expensive, transplant biopsies can result in bleeding from the transplant and even graft loss. In early studies, it has been observed that significant increases in the levels of perforin, granzyme B, and CD3 messenger RNA (mRNA) in urinary cells signal the development of acute transplant rejection. The purpose of this study is to evaluate whether the noninvasive procedure of measuring perforin, granzyme B, and CD3 mRNA levels in urine samples can accurately diagnose and predict kidney transplant rejection, make transplant biopsy unnecessary, and provide an opportunity to initiate treatment for early rejection with the aim to minimize damage to the kidney.

This study will last 3 years post-transplant. There will be a total of 14 study visits. Blood and urine collection will occur at all visits. Additional visits may be necessary for those participants who develop abnormal kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary or redo deceased- or living-donor kidney transplantation
* Ability to provide informed consent

Exclusion Criteria:

* Requires combined organ transplantation
* Previously received a solid organ transplant (other than kidney transplant) or islet cell transplant
* HCV infected
* HIV infected

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have recently undergone kidney transplant
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Shaked, MD, PhD, Study Chair — Department of Surgery, University of Pennsylvania Medical Center; John Friedewald, MD, Principal Investigator — Northwestern University; Stuart Knechtle, MD, Principal Investigator — Department of Surgery, University of Wisconsin; Jean Emond, MD, Principal Investigator — Department of Surgery, Columbia University; Darshana Dadhania, MD, Principal Investigator — Cornell University
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Cornell University, New York, New York
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Dadhania D, Muthukumar T, Ding R, Li B, Hartono C, Serur D, Seshan SV, Sharma VK, Kapur S, Suthanthiran M. Molecular signatures of urinary cells distinguish acute rejection of renal allografts from urinary tract infection. Transplantation. 2003 May 27;75(10):1752-4. doi: 10.1097/01.TP.0000063931.08861.56. PMID 12777869
- [Background] Ding R, Li B, Muthukumar T, Dadhania D, Medeiros M, Hartono C, Serur D, Seshan SV, Sharma VK, Kapur S, Suthanthiran M. CD103 mRNA levels in urinary cells predict acute rejection of renal allografts. Transplantation. 2003 Apr 27;75(8):1307-12. doi: 10.1097/01.TP.0000064210.92444.B5. PMID 12717221
- [Background] Li B, Hartono C, Ding R, Sharma VK, Ramaswamy R, Qian B, Serur D, Mouradian J, Schwartz JE, Suthanthiran M. Noninvasive diagnosis of renal-allograft rejection by measurement of messenger RNA for perforin and granzyme B in urine. N Engl J Med. 2001 Mar 29;344(13):947-54. doi: 10.1056/NEJM200103293441301. PMID 11274620
- [Background] Tatapudi RR, Muthukumar T, Dadhania D, Ding R, Li B, Sharma VK, Lozada-Pastorio E, Seetharamu N, Hartono C, Serur D, Seshan SV, Kapur S, Hancock WW, Suthanthiran M. Noninvasive detection of renal allograft inflammation by measurements of mRNA for IP-10 and CXCR3 in urine. Kidney Int. 2004 Jun;65(6):2390-7. doi: 10.1111/j.1523-1755.2004.00663.x. PMID 15149352
- [Result] Suthanthiran M, Schwartz JE, Ding R, Abecassis M, Dadhania D, Samstein B, Knechtle SJ, Friedewald J, Becker YT, Sharma VK, Williams NM, Chang CS, Hoang C, Muthukumar T, August P, Keslar KS, Fairchild RL, Hricik DE, Heeger PS, Han L, Liu J, Riggs M, Ikle DN, Bridges ND, Shaked A; Clinical Trials in Organ Transplantation 04 (CTOT-04) Study Investigators. Urinary-cell mRNA profile and acute cellular rejection in kidney allografts. N Engl J Med. 2013 Jul 4;369(1):20-31. doi: 10.1056/NEJMoa1215555. PMID 23822777
- See also: Click here for the Clinical Trials in Organ Transplantation [CTOT] public Web site — http://www.ctotstudies.org